CLINICAL TRIAL: NCT04186611
Title: Ergothérapie précoce Aux Soins Intensifs: faisabilité d'implémentation
Brief Title: Early Occupational Therapy in Intensive Care: Feasibility of Implementation
Acronym: ERGO-PRE-SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Marie-Gabrielle Wick Brasey, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ERGO-PRE-SI_2019-00867
Record Dates: First submitted 2019-11-08; First posted 2019-12-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Occupational Therapy; Intensive Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early daily occupational therapy intervention (Experimental): A daily occupational therapy intervention is performed with the patients included. The intervention will consist of assessment as well as early positioning and/or rehabilitation in activities of daily living.
  Interventions: Other: early occupational therapy

INTERVENTIONS:
Other: early occupational therapy — The intervention will be the one usually carried out but earlier and on a daily basis. It will consist of the initial assessment and then positioning and/or carrying out activities of daily living.
  The daily duration of the intervention will be about 45 minutes to 1 hour. The overall duration of the intervention will be determined according to the objectives and will be at most equal to the time of stay in the intensive care unit.

SUMMARY:
The objective of the study is to assess the feasibility of early daily occupational therapy intervention within an interdisciplinary team in an intensive care unit of a Swiss university hospital.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Hospitalized at SMIA for at least 48 hours.
* Stable patient: hemodynamically stabilized patient (norepinephrine dose < 15 mcg/min iv), respiratory (P/F ratio > 150) and neurological (Glasgow Coma Scale > 8).

Exclusion Criteria:

* contraindication to occupational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Early daily occupational therapy intervention feasability (case report form with questions to ask) | Up to intensive care unit discharge, estimated as an average of 6 days
  Assess the feasibility of providing early daily occupational therapy interventions in the Adult Intensive Medicine Service of the Centre Hospitalier Universitaire Vaudois within the current interdisciplinary team. Every day, the occupational therapist complete a case report form which say if the intervention can be realise or not in order to find the feasability of a daily early occupationnal therapy intervention. The feasability is mesure every day for each participant until they leave the intensive care unit.
  the feasibility assessment contains several elements, including the possibility or not of carrying out the intervention, but also the safety aspect with the collection of possible adverse events.

SECONDARY OUTCOMES:
Daily occupational therapy intervention description by completion of case report form | Up to intensive care unit discharge, estimated as an average of 6 days
  Describe the content of the occupational therapy intervention in intensive care unit. Occupational therapists complete a form for each intervention (daily) regarding the type of intervention they have performed with the participants (positioning, daily activities, etc.) until the end of the intervention, when the patient leaves the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland